CLINICAL TRIAL: NCT03076151
Title: Interventional Multicentre Pharmacokinetic Study of Adoport® (Tacrolimus) in Patients With de Novo Kidney Transplantation
Brief Title: Pharmacokinetic Study of Adoport® (Tacrolimus) in Patients With de Novo Kidney Transplantation
Acronym: IMPAKT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I16009 (IMPAKT)
Record Dates: First submitted 2017-02-02; First posted 2017-03-10 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Transplantation; Kidney; Pharmacokinetic
Keywords: Transplantation; Kidney; pharmacokinetic; bayesian estimators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tacrolimus monohydrate (ADOPORT®) (Experimental): patients with de novo Kidney Transplantation under Tacrolimus (ADOPORT®) treatment.
  Interventions: Drug: Tacrolimus monohydrate (ADOPORT®)

INTERVENTIONS:
Drug: Tacrolimus monohydrate (ADOPORT®) — Pharmacokinetic of Tracrolimus (ADOPORT®) on 9 blood sampling by kinetics on 4 kinetics

SUMMARY:
Tacrolimus is a calcineurin inhibitor widely used for the prevention of allograft rejection in solid organ and bone marrow transplantation. It is characterized by a narrow therapeutic index and large inter-individual pharmacokinetic variability. Adoport® is an immediate-release formulation of tacrolimus, to be administered twice daily. Because of a narrow therapeutic window and a better correlation between pre-dose level and effects than between dose and effect, therapeutic drug monitoring (TDM) based on trough whole blood tacrolimus concentrations is recommended for Adoport®. TDM helps to minimize the risk of acute rejection and the occurrence of adverse effects (mainly nephrotoxicity and, to a lesser extent, neurotoxicity).

As reported in a consensus document from a consortium of European experts on tacrolimus TDM, the interdose area-under-the curve (AUC0-12h) is expected to be the best marker of tacrolimus exposure. However, tacrolimus monitoring based on full AUC0-12h is difficult to set up in routine, due to clinical constraints and the necessity of multiple samples. Calculation of the AUC0-12h using Bayesian estimation and a limited sampling strategy, i.e. a few blood samples collected during the early phase post-dose would represent an elegant solution, as already done for other tacrolimus formulations.

Furthermore, the pharmacokinetics (PK) of tacrolimus is influenced by a single nucleotide polymorphism within intron 3 of cytochrome P450 3A5 (CYP3A5). Patients who carry at least one CYP3A5*1 allele are considered to be CYP3A5 expressors (about 12% of the Caucasian population, Hapmap project) and thus require a 1.5 to 2-fold higher starting dose than CYP3A5*3/*3 carriers to reach the predefined target exposure early after transplantation. Although this polymorphism showed no impact on the performance of the Bayesian estimators previously developed for other tacrolimus formulation, the patient status for CYP3A5*3 will be considered in this pharmacokinetic study as a potential covariate in, or confounding factor of, the PK model. Specifically, owing to a 12% frequency in the White European population, about 4 patients carriers of the CYP3A5*1 allele are expected in this study; the performance of the PK model and Bayesian estimator developed will be specifically evaluated in this subgroup.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent of the study
2. Male and female (>= 18 years)
3. Recipients of a first kidney allograft
4. Patients transplanted for less than 7 days at enrolment
5. Patients affiliated to a social security system

Exclusion Criteria:

1. Patients presenting any contraindication to tacrolimus according to the summary of product characteristics of Adoport®
2. Patient presenting anti-HLA antibodies against the graft in pre-transplantation (DSA)
3. Recipients of any transplanted organ other than the kidney
4. Pregnant (positive BHCG test) or lactating women
5. Women without any method of contraception, except for women with no childbearing potential (according to the guidelines of the working group, Clinical Trial Facilitation Group, related to contraception and pregnancy test in clinical trials)
6. Patients participating in any other interventional clinical study at inclusion as well as during the whole course of the current study
7. Patient under judicial protection
8. Patients incapable of understanding the purposes and risks of the study, who cannot give written informed consent, or who are unwilling to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Tacrolimus bayesian estimator performance | Month 3
  The evaluation of Bayesian estimator performance will be based on its capacity to predict tacrolimus AUC (Area Under the Curve), expressed as the bias (%) between the predicted AUC with the PK model and the tacrolimus AUC calculated using the linear trapezoidal rule.

SECONDARY OUTCOMES:
Tacrolimus concentrations predicted by the PK model using a limited sample strategy | Month 3
  The evaluation of the Bayesian estimator performance will be based on its capacity to predict, using a limited number of samples collected during the early phase post-dose, observed tacrolimus AUC0-12h measured using the non-compartmental trapezoidal method with all the time points

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Marquet, MD, Principal Investigator — University Hospital, Limoges
Locations (5):
- France (5):
  - Amiens Picardie University Hospital, Amiens
  - Limoges University Hospital, Limoges
  - Poitiers University Hospital, Poitiers
  - CHU de ROUEN, Rouen
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marquet P, Destere A, Monchaud C, Rerolle JP, Buchler M, Mazouz H, Etienne I, Thierry A, Picard N, Woillard JB, Debord J. Clinical Pharmacokinetics and Bayesian Estimators for the Individual Dose Adjustment of a Generic Formulation of Tacrolimus in Adult Kidney Transplant Recipients. Clin Pharmacokinet. 2021 May;60(5):611-622. doi: 10.1007/s40262-020-00959-y. Epub 2020 Nov 24. PMID 33230714